CLINICAL TRIAL: NCT02005848
Title: Phase II Study to Evaluate the Efficacy and Safety of Human, Alpha-1 Antitrypsin (AAT) [Glassia®] in the Treatment of New Onset Type-1 Diabetes
Brief Title: Phase II Study to Evaluate the Efficacy and Safety of Glassia® in Type-1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kamada-AAT(IV)-011
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: New Onset Type-1 Diabetes
Keywords: Type-1 Diabetes; T1D; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alpha1 Antitrypsin (Glassia) (Experimental): 60 mg/kg body weight
  Interventions: Biological: Alpha-1 Antitrypsin
- Alpha-1 Antitrypsin (Glassia) (Experimental): 120 mg/kg body weight
  Interventions: Biological: Alpha-1 Antitrypsin
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Alpha-1 Antitrypsin
  Other Names: Humman Alpha-1 Antitrypsin; Alpha-1 Proteinase Inhibitor; API; AAT
  Arms: Alpha-1 Antitrypsin (Glassia); Alpha1 Antitrypsin (Glassia)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multicenter, Study Evaluating the Efficacy and Safety of Human, Alpha-1 Antitrypsin (AAT) [Glassia®] in the Treatment of New Onset Type-1 Diabetes.

The study objectives are:

* To assess the efficacy of intravenous AAT in treatment of new onset Type 1 Diabetes
* To assess the safety and tolerability of intravenous AAT in new onset Type 1 Diabetes pediatric and young adult population.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject (or parent/guardian) willing and able to sign an informed consent
* Age 8-25 (inclusive) years
* Recently diagnosed with T1DM
* Basal C-peptide ≥ 0.2 pmol/mL
* Positive for at least one diabetes-related autoantibody
* Ability and consent to comply with completion of patient diary
* No significant abnormalities in serum hematology, serum chemistry
* No significant abnormalities in urinalysis
* No significant abnormalities in ECG
* For women of child bearing potential, non-pregnant, non-lactating female patients

Main Exclusion Criteria:

* IgA deficient subjects
* Subjects who have received an active/ live virus vaccine within 4 weeks of the screening date
* Subjects who have received treatment with corticosteroid medication within 2 months prior to screening or any immunosuppressant or cytostatic agent within 6 months prior to screening
* Individuals with a history of severe immediate hypersensitivity reactions, including anaphylaxis, to plasma products
* Clinically significant intercurrent illnesses
* Pregnant or lactating women
* Current use of any medication known to influence glucose tolerance
* Current or prior (within the last 60 days prior to screening visit) use of metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors or amylin.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2014-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Beta cell function | 12 months from baseline
  Beta cell function (measured by C peptide)

SECONDARY OUTCOMES:
Glycemic control | 12 months from baseline
  Glycemic control expressed in HbA1c level
Beta cell function | 12 months from baseline
Insulin dose | 12 months from baseline
Hypoglycemic episodes | 12 months from baseline
Safety parameters | 12 months from baseline
  Adverse events, vital signs, physical examination

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Schneider Children's Medical Center, Pethach Tikva
  - Assaf Harofe Medical Center, Ẕerifin